CLINICAL TRIAL: NCT04128384
Title: Changes in Infranodal Conduction Times and New Onset Left Bundle Branch Block: Possible Predictors for High-grade AV Block Following Transcatheter Aortic Valve Replacement
Brief Title: Infranodal Conduction Time During TAVR as Predictor of HAVB
Acronym: HOM-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Christian Ukena, Principal Investigator, University Hospital, Saarland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HOM-TAVI
Record Dates: First submitted 2019-10-12; First posted 2019-10-16 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Severe Aortic Valve Stenosis; High-degree AV Block; Left Bundle-Branch Block
Keywords: Transcatheter valve replacement; Infranodal conduction time; High-degree AV block; Left Bundle-Branch Block
MeSH Terms: conditions — Aortic Valve Stenosis; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EPS arm (Other): Limited electrophysiologic study including measurements of HV- and AH-intervals pre- and post-TAVR
  Interventions: Diagnostic Test: Limited electrophysiologic study including measurements of HV- and AH-intervals pre- and post-TAVR

INTERVENTIONS:
Diagnostic Test: Limited electrophysiologic study including measurements of HV- and AH-intervals pre- and post-TAVR — For the purpose of obtaining intracardiac measurements, the quadripolar diagnostic catheter used as temporary pacemaker wire (5F, Woven, Boston Scientific) during TAVR was retracted from the apex and positioned at the His bundle to measure HV- and AH-intervals.

SUMMARY:
Consecutive patients with high grade aortic stenosis undergoing transcatheter aortic valve replacement (TAVR) with a self-expanding valve (Medtronic CoreValve Evolut R® or Edwards Sapien S3®) without pre-existing pacemaker devices are eligible for inclusion. During the TAVR procedure, an electrophysiologic study including measurements of infranodal conduction times (HV-interval before and after valve implantation) will be performed. Electrocardiograms before TAVR, before discharge, after 30 days and after 12 months will be analyzed regarding new onset LBB and the occurrence of high-degree AV block (HAVB) .

ELIGIBILITY:
Inclusion Criteria:

1. Indication for TAVR according to current guidelines
2. Written informed consent

Exclusion Criteria:

1. Pre-existent intracardiac device as pacemaker, implanted cardioverter defibrillator or CRT-P/CRT-D device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
High-degree AV block | 24 months
  Occurence of high-degree AV block necessitating a pacemaker implantation during follow up
Persistence of left bundle-branch block | 24 months
  Persistence of new onset left bundle branch-block following TAVR procedure

SECONDARY OUTCOMES:
Differences between implanted valve types on ifranodal conduction | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ukena, MD, Principal Investigator — Universitätsklinikum des Saarlandes, Homburg/Saar, Germany
Locations (1):
- Universitätsklinikum des Saarlandes, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaede L, Kim WK, Liebetrau C, Dorr O, Sperzel J, Blumenstein J, Berkowitsch A, Walther T, Hamm C, Elsasser A, Nef H, Mollmann H. Pacemaker implantation after TAVI: predictors of AV block persistence. Clin Res Cardiol. 2018 Jan;107(1):60-69. doi: 10.1007/s00392-017-1158-2. Epub 2017 Sep 29. PMID 28963581
- [Background] Nazif TM, Williams MR, Hahn RT, Kapadia S, Babaliaros V, Rodes-Cabau J, Szeto WY, Jilaihawi H, Fearon WF, Dvir D, Dewey TM, Makkar RR, Xu K, Dizon JM, Smith CR, Leon MB, Kodali SK. Clinical implications of new-onset left bundle branch block after transcatheter aortic valve replacement: analysis of the PARTNER experience. Eur Heart J. 2014 Jun 21;35(24):1599-607. doi: 10.1093/eurheartj/eht376. Epub 2013 Oct 30. PMID 24179072
- [Background] Urena M, Mok M, Serra V, Dumont E, Nombela-Franco L, DeLarochelliere R, Doyle D, Igual A, Larose E, Amat-Santos I, Cote M, Cuellar H, Pibarot P, de Jaegere P, Philippon F, Garcia del Blanco B, Rodes-Cabau J. Predictive factors and long-term clinical consequences of persistent left bundle branch block following transcatheter aortic valve implantation with a balloon-expandable valve. J Am Coll Cardiol. 2012 Oct 30;60(18):1743-52. doi: 10.1016/j.jacc.2012.07.035. Epub 2012 Oct 3. PMID 23040577
- [Derived] Pavlicek V, Mahfoud F, Bubel K, Fries P, Ewen S, Bohm M, Scheller B, Ukena C. Prediction of conduction disturbances in patients undergoing transcatheter aortic valve replacement. Clin Res Cardiol. 2023 May;112(5):677-690. doi: 10.1007/s00392-023-02160-0. Epub 2023 Jan 21. PMID 36680617